CLINICAL TRIAL: NCT00152958
Title: A Double-blind, Placebo-controlled, Randomised Withdrawal Study of 3 Month Duration in Patients Suffering From Idiopathic Restless Legs Syndrome Who Responded to a Preceding, 6-month Treatment With Open-label Pramipexole Including Titration (0.125, 0.25, 0.5, 0.75 mg Orally q.n.)
Brief Title: A Study in Patients Suffering From Idiopathic Restless Legs Syndrome Who Responded to a Preceding, 6-month Treatment With Open-label Pramipexole Including Titration (0.125, 0.25, 0.5, 0.75 mg Orally q.n.)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 248.546
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole

INTERVENTIONS:
Drug: Pramipexole

SUMMARY:
The primary objective is to assess sustained efficacy in patients who have responded to a 6 month treatment with open-label pramipexole.

Secondary objectives are the measurement of severity of the RLS, assessment of early withdrawal phenomena after termination of trial medication, augmentation under treatment, sleepiness, quality of life and subjective wellbeing, the physician's clinical assessment of symptom severity and improvement. Another secondary objective is safety and tolerability of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female out-patients aged 18-80
* Diagnosis of idiopathic RLS according to the Clinical RLS criteria of the International RLS Study Group
* RLSRS score > 15
* RLS symptoms present at least 2 to 3 days per week within the last 3 months
* Written informed consent

Exclusion Criteria:

* Women of childbearing potential without adequate contraception, or breastfeeding
* Concomitant or previous pharmacologically therapy of RLS
* Clinically significant renal disease, and/or hepatic disease
* Any of the following lab results at screening: Hb, TSH, T3 or T4, clinically significantly out of normal range, positive urine drug screen
* Other clinically significant metabolic-endocrine (including diabetes mellitus requiring insulin therapy), haematological, gastro-intestinal disease or pulmonary disease . Poorly controlled cardiovascular disease
* History or clinical signs of peripheral neuropathy (PNP), myelopathy or multiple sclerosis or any other neurological disease, with potential to secondarily cause RLS symptoms, history of or clinical signs for any form of epilepsy or seizures
* Presence of any sleep disorder
* History of schizophrenia or any psychotic disorder, history of mental disorders, alcohol abuse or drug addiction
* History of or clinical signs of malign neoplasm
* Patients on a shift-work-schedule, or who are otherwise unable to follow a regular sleep-wake cycle enabling use of study medication at times indicated
* Allergic to pramipexole or its excipients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224
Dates: Start 2004-01; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Time to target event (CGI-I rating in association with RLSRS score above 15, period 2) for full analysis set | from randomization up to 3 months

SECONDARY OUTCOMES:
Time to target event for per protocol set (period 2) | from randomization up to 3 months
Number of target events (period 2) | from randomization up to 3 months
Change from baseline (visit 10) in the total score of Restless Legs Syndrome Rating Scale for Severity (RLSRS) (period 2) | from randomization up to 3 months
Clinical Global Impressions - Global Improvement (period 2) | from randomization up to 3 months
Change from baseline (visit 10) in Clinical Global Impressions - Severity of illness score (CGI-S) by 2 or more categories (period 2) | from randomization up to 3 months
Clinical Global Impressions - Therapeutic Effect (CGI-TE) (period 2) | from randomization up to 3 months
Clinical Global Impressions - Side Effects (CGI-SE) (period 2) | from randomization up to 3 months
Change in Patient global impression (PGI) (period 2) | from randomization up to 3 months
Change from baseline (visit 10) in Johns Hopkins Quality of Life (RLS-QoL) score (period 2) | from randomization up to 3 months
Change from baseline (visit 10) in Visual analogue scales (RLS-VASs) for assessment of RLS symptoms (period 2) | from randomization up to 3 months
Change from baseline (visit 10) in Epworth sleepiness scale (ESS) | from randomization up to 3 months
Change from baseline (visit 2) in Augmentation severity rating scale of IRLSSG (ASRS) (period 2) | up to 9 months
Change from baseline ASRS (period 1) | up to 6 months
Change from baseline in the total score of RLSRS (period 1) | up to 6 months
RLSRS responder status by visit (non-responder, partial responder, responder) (period 1) | after 6 months
RLSRS responder status for patients who discontinued the study prematurely in period 1 by reason for discontinuation (period 1) | up to 6 months
Clinical Global Impressions - Global Improvement (period 1) | 6 months
Clinical Global Impressions - Severity of illness score (CGI-S) (period 1) | 6 months
Clinical Global Impressions - Therapeutic Effect (CGI-TE) (period 1) | 6 months
Clinical Global Impressions - Side Effects (CGI-TE) (period 1) | 6 months
Change in patient global impression from baseline (period 1) | 6 months
Change from baseline in Johns Hopkins Quality of Life (RLS-QoL) score (period 1) | 6 months
Change from baseline in RLS-VASs (period 1) | 6 months
Change from baseline in ESS | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (12):
- Germany (12):
  - Boehringer Ingelheim Investigational Site, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - emovis GmbH, Berlin
  - Boehringer Ingelheim Investigational Site, Chemnitz
  - ClinPharm Internat. GmbH & Co. KG, Görlitz
  - Clinpharm International GmbH & Co. KG, Hellersdorf
  - Paracelsus-Elena-Klinik, Kassel
  - ClinPharm International GmbH & Co. KG, Leipzig
  - Neurologische Klinik der Otto-von-Guericke-Universität, Magdeburg
  - Universitätsklinikum Giessen und Marburg, Marburg
  - Boehringer Ingelheim Investigational Site, München
  - Boehringer Ingelheim Investigational Site, Würzburg